CLINICAL TRIAL: NCT00331721
Title: A Multicentre, Double-Blind, Randomised, Placebo-Controlled, Dose-Escalating Parallel-Group Study to Investigate the Tolerability of Enecadin (INN) in Acute Ischemic Stroke
Brief Title: Tolerability of Enecadin (INN) in Acute Ischemic Stroke Trial - TEST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Scientific data called into question the viability of the substance class
Sponsor: PAION Deutschland GmbH (Industry)
Responsible Party: Karin Wilhelm-Ogunbiyi, MD / Medical Director & Head of Clinical Development, PAION Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PN06-CLD-01001
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Stroke
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Enecadin
  Interventions: Drug: Enecadin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enecadin — Dose escalating
  Arms: 1
Drug: Placebo — Placebo comparator
  Arms: 2

SUMMARY:
The main objective of this study is to investigate the tolerability of enecadin in patients with acute ischemic stroke. Furthermore, the pharmacokinetics of enecadin in both male and female patients with acute ischemic stroke will be assessed. Efficacy trends will be evaluated up to day 30 post stroke.

DETAILED DESCRIPTION:
In the acute stage of ischemic stroke, an ischemic core characterized by a marked decrease in blood flow is present, leading to irreversible neuronal damage at an early stage. Around the boundary of the ischemic core, there is a region called ischemic penumbra in which functional recovery is possible after recirculation of blood flow within several hours after the onset, even though the blood flow is markedly decreased. Prevention of nerve cell death in the ischemic penumbra by neuroprotective therapy should greatly improve outcome and prognosis of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke (scoring 3-20 on the National Institutes of Health Stroke Scale [NIHSS]) with level of consciousness score: 0 or 1 (conscious patients) are eligible to be treated within 9 hours of onset of stroke symptoms.
* For female patients: post-menopausal or surgically sterile (post-menopausal: age ≥55 years and last menses ≥3 years ago).

Exclusion Criteria:

* Participation in any investigational study in the previous 30 days.
* Patients unable to understand trial related information.
* History or evidence of severe heart diseases further specified in the protocol.
* History or evidence of additional diseases or results of baseline visit as specified in the protocol.
* Use of concomitant and prior medications as defined in the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Safety parameters, Pharmacokinetics & trends of efficacy | One month

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Ringleb, Dr., Principal Investigator — Heidelberg University
Locations (26):
- Austria (2):
  - Investigational Site 1, Linz
  - Investigational Site 2, Linz
- Belgium (3):
  - Investigational Site, Antwerp
  - Investigational Site, Bruges
  - Investigational Site, Leuven
- Germany (21):
  - Investigational Site, Aachen
  - Investigational Site, Bad Neustadt an der Saale
  - Investigational Site, Bergisch Gladbach
  - Investigational Site, Berlin
  - Investigational Site, Bochum
  - Investigational Site, Dortmund
  - Investigational Site, Dresden
  - Investigational Site, Erlangen
  - Investigational Site, Frankfurt
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Hamburg
  - Investigational Site, Hanover
  - University of Heidelberg, Heidelberg
  - Investigational Site, Ingolstadt
  - Investigational Site, Leipzig
  - Investigational Site, Magdeburg
  - Investigational Site, Minden
  - Investigational Site, Munich
  - Investigational Site, Nuremberg
  - Investigational Site, Remscheid
  - Investigational Site, Wiesbaden